CLINICAL TRIAL: NCT01065623
Title: An Open Label Phase I Dose-escalation Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Maximum Tolerated Dose of BAY79-4620 Administered as an Intravenous Infusion Once Every 2 Weeks in Patients With Advanced Solid Tumors
Brief Title: Clinical Study to Evaluate the Maximum Tolerated Dose of BAY79-4620 Given Every 2 Weeks to Patients With Advanced Solid Tumors
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The study was terminated due to safety reasons
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12672; 2009-015085-58 (EudraCT Number)
Record Dates: First submitted 2010-02-08; First posted 2010-02-09 (Estimated); Last update posted 2014-10-01 (Estimated); Status verified 2014-09

CONDITIONS: Neoplasms
Keywords: Phase I; Dose escalation; Immunoconjugate
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Experimental)
  Interventions: Drug: BAY79-4620

INTERVENTIONS:
Drug: BAY79-4620 — 1-hour infusion every 14 days. Starting dose will be 0.15 mg/ kg and dose will be escalated dependent on any dose limiting toxicities

SUMMARY:
Clinical study to determine safety, tolerability, to measure how the drug is metabolized by the body and to determine the maximum tolerated dose of BAY79-4620 given every 2 weeks to patients with advanced solid tumors

ELIGIBILITY:
Inclusion Criteria:

* The informed consent must be signed before any study specific tests or procedures are done
* Male or female patients aged >18 years
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 - 2
* Life expectancy of at least 12 weeks
* Patients with advanced, histologically or cytologically confirmed solid tumors, refractory to any standard therapy, have no standard therapy available, or patients must have actively refused any treatment which would be regarded standard, and/or if in the judgment of the investigator or his designated associate(s), experimental treatment is clinically and ethically acceptable
* Radiographically or clinically evaluable tumor
* Adequate bone marrow, liver, and renal functions as assessed by the following laboratory requirements to be conducted within 14 days prior to start of first dose

Exclusion Criteria:

* History of cardiac disease: congestive heart failure (CHF) > NYHA Class II; myocardial infarction within 3 months prior to study entry; new onset angina within 3 months or unstable angina or cardiac arrhythmias requiring anti-arrhythmic therapy (beta blockers or digoxin are permitted)
* Uncontrolled hypertension defined as systolic blood pressure >160 mmHg and/or diastolic blood pressure >95 mmHg, despite optimal medical management
* Symptomatic metastatic brain or meningeal tumors unless the patient is >6 months from definitive therapy, has no evidence of tumor growth on an imaging study within 2 weeks prior to study entry, and is clinically stable with respect to the tumor at the time of study entry.
* Patients with severe renal impairment or on dialysis
* Known human immunodeficiency virus (HIV) infection or patients with an active hepatitis B or C infection necessitating treatment. Patients with chronic hepatitis B or C are eligible
* Active clinically serious infections of Common Terminology Criteria for Adverse Events Version 3 (CTCAE v3.0) > Grade 2
* Serious, non-healing wound, ulcer, or bone fracture
* Major surgery, open biopsy, or significant trauma within 4 weeks prior to the first dose of study drug
* Anticancer chemotherapy, experimental cancer therapy, or immunotherapy within 2 weeks of start of first dose
* Radiotherapy to the target lesions within 3 weeks prior to Cycle 1 Day 1 (first dose of study drug). Palliative radiotherapy will be allowed as described in the study protocol. Radiotherapy to the target lesions during study will be regarded as progressive disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2010-04; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Adverse Event reporting | Approximately 3 years after initiation of the trial
Pharmacokinetics profile of BAY79-4620 | End of cycle 2 (14 days per cycle)

SECONDARY OUTCOMES:
Biomarkers evaluation | Approximately 3 years after initiation of the trial
Tumor response evaluation | Approximately 3 years after initiation of the trial
Immunogenicity evaluation | Approximately 3 years after initiation of the trial

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (2):
- Netherlands (2):
  - Rotterdam
  - Utrecht